CLINICAL TRIAL: NCT02935140
Title: Safe Use of Speaking Valve in Children During Sleep Using Trans-tracheal Pressure Measurement
Status: Completed | Type: Observational
Sponsor: St Mary's Hospital for Children (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-09
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Lung Disease of Prematurity; Chronic Respiratory Failure
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Many children who are born medically fragile due to prematurity, multiple congenital abnormalities or an acquired insult (i.e. cardiac, neurologic, etc.) may require tracheostomy tube placement due to need of chronic respiratory support. Patients on tracheostomy tubes are often unable to vocalize, causing a delay in speech development and poor speech. To help restore normal phonation and promote language development in young pediatric patients with tracheostomies, speaking valves are used. Previously it was shown that the Passy-Muir speaking valve was safe to use during sleep in children by showing there were no adverse cardiopulmonary events seen. One objective measurement that was not evaluated was trans-tracheal pressure manometry. The purpose of this study is to continue to validate the safety of the Passy-Muir speaking valve while asleep, with the use of trans-tracheal manometry by comparing expiratory pressure manometry while the patient is awake and asleep.

DETAILED DESCRIPTION:
Previously it was shown that the Passy-Muir speaking valve was safe to use during sleep in children. There were no adverse cardiopulmonary events seen while wearing the speaking valve during sleep. However, trans-tracheal pressure was not measured while these children were asleep wearing the Passy-Muir speaking valve.The investigators hypothesize that patients who tolerate speaking valve while awake will have similar trans-tracheal pressure measurement when asleep as when they are awake.

The specific aims of this proposal are:

1) to show that the Passy-Muir speaking valve worn during sleep has similar trans-tracheal pressure manometry as when worn while awake.

The primary outcome measure is to show that trans-tracheal manometry measurement is similar while on the Passy-Muir speaking valve when patients are awake and asleep

Secondary outcomes are a) recording of symptoms (i.e. choking, gagging, increased respiratory rate, abnormal breathing pattern, coughing, chest tightness and aversion) while wearing the speaking valve either awake or asleep b) recording vital signs which will be compared to normal and baseline for age (i.e. heart rate, respiratory rate, end-tidal carbon dioxide and oxygen saturation) while awake and asleep.

Background and significance:

Previously it was shown that Passy-Muir speaking valve is safe to use during sleep in children. However it continues to be contraindicated for use while asleep. A small prospective study done on 10 tracheostomized adult patients with a mean age of 70 years showed that the use of the speaking valve for one night in seriously ill patients was not associated with apneas or significant desaturations. A cohort study of 32 tracheostomized patients showed that 14 patients were able to tolerate speaking valve for 24 hours; even during sleep.

Pediatric patients with tracheostomy tube are often unable to vocalize. Tracheostomy tubes allow the exhaled flow of air to bypass the vocal cords out through the opening of the tube making speech difficult. This causes a delay in speech development and poor speech. Speaking valves, like the Passy-Muir valve, restore normal phonation and promote language development in young pediatric patients with tracheostomies. Speech development is not the only benefit seen with speaking valves. Speaking valves can lead to improvement in swallowing safety reducing aspiration, improved ventilator weaning leading to more rapid tracheal decannulation, reduce secretion management, improve hygiene, and enhance smell and taste.

Evaluation of speaking valve tolerance can be done by monitoring vital signs (i.e. respiratory rate, heart rate, and oxygen saturation). In addition, measurement of trans-tracheal pressure is an invaluable tool in evaluating subjects for speaking valve placement. Measurement of trans-tracheal pressure is predictive of good tolerance of the valve.

The measurement allows one to quickly and easily assess patency of the upper airway and the ability to force air through the vocal cords. If the pressures are elevated, greater than 10 cm of water on inhalation phase and 30cm of water on the exhalation phase, it would indicate an obstruction in the upper part of the trachea (i.e. subglottic stenosis). The pressures can also evaluate respiratory function prior to considering patients for placement of the valve.

Many children who are born medically fragile due to prematurity, multiple congenital abnormalities or an acquired insult (i.e. cardiac, neurologic, etc.) may require tracheostomy tube placement due to need of chronic respiratory support. Initially, after a patient is assessed for a speaking valve and is cleared for use, a patient may be apprehensive toward the speaking valve.

If a patient displays discomfort, anxiety, dyspnea/respiratory distress or there is air trapping (from the build-up of subglottic pressure from incomplete exhalation) trials are repeated on subsequent days. However, one can assume that initial failure is due to aversion, but it may be due to resistance in the upper airway, or vice versa.

The purpose of this study is to continue to validate the safety of the Passy-Muir speaking valve while asleep, with the use of trans-tracheal manometry by comparing expiratory pressure manometry while the patient is awake and asleep.

ELIGIBILITY:
Inclusion Criteria:

i. Any subject between the ages of 0-18 years of age who is a resident of St Mary's Healthcare System for Children with a chronic tracheostomy may be enrolled. Patients have to be approved for a Passy-Muir speaking valve as per St Mary's Healthcare System for Children written policy.

Exclusion Criteria:

i. Patients who do not meet the criteria for the use of speaking valve (i.e. unconscious and/or comatose patients, patients who require 24-hour inflated tracheostomy tube cuff due to inadequate ventilation, foam-filled tracheostomy tube, severe airway obstruction, unmanageable thick secretions, severe risk for aspiration, severely reduced lung elasticity, and not intended for use with endotracheal tubes).

ii. Patients with an acute illness and is not at baseline status. iii. Have any kind of respiratory distress.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Number of Subjects: The current number of subjects at St Mary's Healthcare System for Children approved and tolerates the Passy-Muir speaking valve are eight. All eight children will be recruited for the study.
  Gender of Subjects: Both males and females subjects will be eligible for this study
  Age of Subjects: Children ages 0-18 yrs old.
  Racial and Ethnic Origin: All races and ethnic origins will be eligible for this study
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Trans-tracheal Pressure Measurement | one day
  trans-tracheal manometry measurement is similar while on the Passy-Muir speaking valve when patients are awake and asleep

SECONDARY OUTCOMES:
Recording of symptoms | one day
  a) recording of symptoms (i.e. choking, gagging, increased respiratory rate, abnormal breathing pattern, coughing, chest tightness and aversion) while wearing the speaking valve either awake or asleep
vital signs | one day
  b) recording vital signs which will be compared to normal and baseline for age (i.e. heart rate, respiratory rate, end-tidal carbon dioxide and oxygen saturation) while awake and asleep.

CONTACTS AND LOCATIONS:
Overall Officials: Melodi Pirzada, MD, Principal Investigator — St Mary's Healthcare System for Children

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Barraza GY, Fernandez C, Halaby C, Ambrosio S, Simpser EF, Pirzada MB, Islam S. The safety of tracheostomy speaking valve use during sleep in children: a pilot study. Am J Otolaryngol. 2014 Sep-Oct;35(5):636-40. doi: 10.1016/j.amjoto.2014.04.011. Epub 2014 May 4. PMID 24888795
- [Result] Brigger MT, Hartnick CJ. Drilling speaking valves: a modification to improve vocalization in tracheostomy dependent children. Laryngoscope. 2009 Jan;119(1):176-9. doi: 10.1002/lary.20077. PMID 19117281
- [Result] Buckland A, Jackson L, Ilich T, Lipscombe J, Jones G, Vijayasekaran S. Drilling speaking valves to promote phonation in tracheostomy-dependent children. Laryngoscope. 2012 Oct;122(10):2316-22. doi: 10.1002/lary.23436. Epub 2012 Jul 9. PMID 22777746
- [Result] Hopkins C, Whetstone S, Foster T, Blaney S, Morrison G. The impact of paediatric tracheostomy on both patient and parent. Int J Pediatr Otorhinolaryngol. 2009 Jan;73(1):15-20. doi: 10.1016/j.ijporl.2008.09.010. Epub 2008 Nov 18. PMID 19019462
- [Result] Johnson DC, Campbell SL, Rabkin JD. Tracheostomy tube manometry: evaluation of speaking valves, capping and need for downsizing. Clin Respir J. 2009 Jan;3(1):8-14. doi: 10.1111/j.1752-699X.2008.00100.x. PMID 20298366